CLINICAL TRIAL: NCT05137353
Title: RitMoZ Training: A Randomized Control Trial Study to Assess a Multisensory Music Intervention for Children With Reading Disorders in Hungary
Brief Title: A Multisensory Music Intervention for Children With Reading Disorders (RitMoZ)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Centre for Natural Sciences (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, Ferenc Honbolygo, PhD, Senior Research Fellow, Research Centre for Natural Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-Prism-C ESR-10 project; H2020-MSCA-ITN-2018 813546 (Other Grant/Funding Number: MARIE SKŁODOWSKA-CURIE INNOVATIVE TRAINING NETWORK (ITN))
Record Dates: First submitted 2021-11-28; First posted 2021-11-30 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Reading Disorder
Keywords: reading disorders; music intervention; rhythmic stimulations; phonological processing; Event-Related Brain Potentials
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Training (RitMoZ Training) (Experimental): 12 sessions spread in the course of 1.5 months: each session has a duration of 90 minutes; each week will have 2 sessions
  Interventions: Behavioral: Music Training (RitMoZ Training)
- Spelling Training (Active Comparator): 12 sessions spread in the course of 1.5 months: each session has a duration of 90 minutes; each week will have 2 sessions
  Interventions: Behavioral: Spelling Training

INTERVENTIONS:
Behavioral: Music Training (RitMoZ Training) — This training is inspired by intervention concepts followed in SUVAG Polyclinic in Zagreb, Croatia and Kodaly pedagogy in Hungary. RitMoZ Training programme consists of 6 main activities: matching activity, nursery rhymes, rhythmic stimulations, music shapes, music writing and music reading. The training focuses on the perceptual overlap between language and music, embodiment and entrainment. The aim of the training is to improve characteristic features of reading disorders such as phonological awareness, perception of rhythm, phonological working memory and perception of speech sounds.
  Arms: Music Training (RitMoZ Training)
Behavioral: Spelling Training — This training consists of activities which focus on practicing spelling words in a computer task; the aim is to train orthographic processing which is suggested to improve phonological awareness and phonological working memory.
  Arms: Spelling Training

SUMMARY:
With this study, we wish to test how effective/ beneficial music activities can be for children with dyslexia.

DETAILED DESCRIPTION:
Studies have shown that music in the form of training (i.e., intervention) is able to facilitate linguistic processes (e.g., phonological encoding/decoding, categorical perception) and cognitive functions (e.g., working memory) in children that have dyslexia or reading difficulties. In addition to this, music trainings with a focus on entrainment can improve phonological as well as reading skills.

In line with the above, we have designed and developed a music training programme. This programme, which is called RitMoZ Training (i.e., from Ritmus és Mozgás és Zene: meaning Rhythm and Movement and Music in Hungarian language), is designed for (Hungarian) children who have dyslexia or reading difficulties.

In order to assess the efficacy of the music training, we are going to conduct a randomized controlled trial which consists of a pre-training phase, a training phase and a post-training phase.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of reading disorder
* Hungarian as native language

Exclusion Criteria:

* comorbidities (e.g., Attention Deficit Disorder (ADD), Attention Deficit Hyperactivity Disorder (ADHD))
* sensory impairment (e.g., hearing loss, low vision)
* cognitive impairment (e.g., panic disorder, low IQ)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Reading test | 4 minutes
  For the assessment of the ability to read aloud series of high frequency words, low frequency words and pseudowords, is applied from the shortened 3DM-H (Differential Diagnostics of Dyslexia Maastricht - Hungarian adaptation). With this test, reading speed, fluency and accuracy and pseudoword accuracy are measured.
Spelling test | 4-7 minutes
  For the assessment of spelling, the present subtest is applied from the shortened version of the 3DM-H. Both spelling accuracy and reaction time are measured.
Phoneme deletion test | 3-7 minutes
  For the assessment of phoneme deletion, the present subtest is applied from the shortened version of the 3DM-H. Both accuracy and reaction time are measured.
Letter-sound identification test | 2-3 minutes
  For the assessment of letter-sound identification, the present subtest is applied from the shortened version of the 3DM-H. Both accuracy and reaction time are measured.
Letter-sound discrimination test | 2 - 4 minutes
  For the assessment of letter-sound discrimination, the present subtest is applied from the shortened version of the 3DM-H. Both accuracy and reaction time are measured.
Rapid Automatized Naming (RAN) test | 3-5 minutes
  To assess rapid naming of letters, digits and objects, the present subtest is applied from the shortened version of the 3DM-H. Here, the processing speed is measured.
Choice reaction time test | 1 - 2 minutes
  The present subtest is applied from the shortened version of the 3DM-H; here, the reaction time is measured.
Lexical decision task | 12- 15 minutes
  To assess lexical decision, the present test is applied. Here, accuracy is measured.
Auditory discrimination of acoustic and phonetic alteration of pseudowords | 20 minutes
  This is an Event-Related Potentials (ERPs) task where a speech multifeature paradigm is applied. In the current task, the amplitudes of the Mismatch Negativity (MMN) responses - which are elicited in certain time windows - are measured in every condition.

CONTACTS AND LOCATIONS:
Overall Officials: Ferenc Honbolygó, PhD, Principal Investigator — Research Centre for Natural Sciences
Locations (1):
- Research Centre for Natural Sciences, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This is the website which provides information and details about the intervention and the study procedure. — https://www.ritmozintervention.com/